CLINICAL TRIAL: NCT04290364
Title: Early Palliative Care for Patients With Pancreatic Cancer - Health Care Service Use and Quality of Life - a Quasi-experimental Study Using Historical Controls
Brief Title: Early Palliative Care in Pancreatic Cancer - a Quasi-experimental Study
Acronym: PanEffort-1
Status: Completed | Type: Observational
Sponsor: Inge Høgh Dufva (Other)
Responsible Party: Sponsor-Investigator, Inge Høgh Dufva, Consultant, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Other Study IDs: PanEffort-1
Record Dates: First submitted 2020-02-20; First posted 2020-02-28 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
Keywords: Palliative care
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Patients newly diagnosed with pancreatic cancer included in the prospective part of the study
  Interventions: Other: Palliative care
- Retrospective cohort: Patients diagnosed with pancreatic cancer before early palliative care was introduced (historical control patients)

INTERVENTIONS:
Other: Palliative care — The patients in the prospective part of the study are seen on home-visits and offered standard palliative care within three weeks of diagnosis.
  Groups: Prospective cohort

SUMMARY:
The aim of the proposed study is to understand the palliative care needs of patients with pancreatic cancer, to investigate whether early palliative care can improve patient outcomes and reduce use of health care services, and to understand the psychological health of carers and their satisfaction with care.

A quasi-experimental design is used, introducing palliative care for patients with pancreatic cancer within three weeks from diagnosis. The patients are recruited in Dept. of Surgery, Hospital of North Zealand, which covers the northern catchment area of the Capital Region of Copenhagen, Denmark. Patients are seen by the palliative care team on home-visits every four weeks throughout their trajectory, and quality of life is evaluated using the following quality of life questionnaires (QLQs): European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients receiving palliative care (EORTC QLQ-C15-PAL), European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Pancreatic Cancer Patients (EORTC QLQ-PAN26), and Hospital Anxiety and Depression Scale (HADS). For carers, mental health is evaluated using HADS and satisfaction with care is evaluated using the Family Caregivers' Satisfaction With Palliative Care in Advanced Cancer Questionnaire (FAMCARE-2).

The primary outcome is health care service use (acute hospital admissions, days in hospital). Secondary outcomes are survival and place of death. Data are compared with historical control patients treated in the same hospital before introduction of early palliative care. These outcomes are readily available from patient records and are expected to carry a very low risk of bias.

Palliative care needs at referral in the study group will be compared with palliative care needs in the subgroup of historical control patients referred to palliative care on-demand.

For outcomes where unbiased historical control data are not available a prospective observational approach is used. These include symptom burden, weight, psychological health and satisfaction with care.

The minimum sample size needed to show a clinically significant decrease in acute hospital admissions is 70, 35 participating in the prospective study and 35 historical control patients. The study will include 40-50 patients and their carers from September 2019 to September 2020.

DETAILED DESCRIPTION:
Study design

All patients with symptoms compatible with pancreatic cancer living in the northern catchment area of the Capital Region of Copenhagen, Denmark, are referred to Dept. of Surgery, Hospital of North Zealand for further investigations. Cases diagnosed with pancreatic cancer are discussed at a regional Multi-Disciplinary-Team (MDT) conference and either referred for surgery or chemotherapy or receive best supportive care in Dept. of Surgery. The Palliative Care Unit at Hospital of North Zealand covers the same geographical area with 310,000 inhabitants.

Patients referred to Dept. of Surgery and diagnosed with pancreatic cancer are offered participation in this study. All participants will receive home-visits from the palliative care team every four weeks, starting within three weeks from diagnosis and until end-of-life or cure without residual palliative needs.

The study design chosen is a quasi-experimental design using historical control patients for the primary outcome: use of health care services (acute hospital admissions, days in hospital) and the secondary outcomes: survival and place of death. The historical control patients were diagnosed before the introduction of early palliative care. The outcomes are readily available from patient records and are expected to carry a very low risk of registration bias. Palliative care needs at referral in the study group will be compared with palliative care needs in the subgroup of historical control patients referred to palliative care on-demand.

Demographic data will be collected for participants and historical controls to evaluate if any selection bias or other systematic differences exist between the groups.

For outcomes where unbiased historical control data are not available a prospective observational approach is used. These include symptom burden, psychological health and satisfaction with care.

The study will include 40-50 patients and their carers from September 2019 to September 2020.

Amendment 19th Nov. 2020: The number of patients and carers included increased to 70-75 to allow for subgroup analyses.

Recruitment and informed consent

Recruitment to this project will take place in Dept. of Surgery, Hospital of North Zealand to which all patients suspected of having pancreatic cancer and living in the northern catchment area of the Capital Region of Copenhagen will be referred for further investigations. The patients will be informed about their diagnosis by the responsible surgeon in the outpatient clinic in an undisturbed environment. The patients will then be informed about the possibility of participation in the present study. They will receive both oral and written information about the project and will be allowed enough time to consider participation before deciding, as long as it allows contact to the palliative care team within three weeks from diagnosis. It is expected that most patients will come to Dept. of Surgery with a family member or friend, as they are aware that they will receive the results from the investigations performed. However, patients will be informed that they have a right to come back for further information about the protocol accompanied by a family member or any other person they want to bring. They will meet either a surgeon or a palliative care physician who can give further information and answer any possible questions at this meeting.

Written informed consent will be obtained before any protocol related procedures are performed.

Carers will receive separate oral and written information either on the same day as the patient or when meeting the palliative care team on the first visit. Carers will sign a separate consent form if they want to participate in the study. Carers have the same rights as the patients regarding time for consideration and further information before signing the consent form.

Palliative Care Intervention

Patients and carers will be seen on home-visits. The first time they will meet a doctor and usually also a nurse, while follow-up home-visits can be undertaken by either a doctor or a nurse. Home-visits are scheduled every four weeks. Patients can contact a doctor or a specialised nurse on weekdays for consultation. The palliative care nurse will contact a palliative care physician if needed for change of treatment or other reasons. Palliative care is offered in parallel with any specific cancer treatment given.

The patients will receive standard palliative care including treatment of symptoms (e.g. pain, nausea, weight loss, loss of appetite, diarrhoea or fatigue), psychosocial support, physiotherapy, nutritional counselling and advance care planning, depending on their needs. The palliative care team comprises physicians, nurses, a physiotherapist and a chaplain. Patients and/or carers scoring 8 or more on HADS for anxiety and/or depression will be advised to be referred to a psychologist via their general practitioner.

Change from standard of care

Patients with pancreatic cancer are normally referred to palliative care when the surgeon, oncologist or general practitioner taking care of them find that they are not able to meet their palliative care needs, or if the patients and their families request a referral. Most patients are referred late in their trajectory and only half of the patients are referred. We do not know whether patients not referred to palliative care in the routine setting have palliative care needs, whether they are met by other physicians or whether they have unsolved palliative care needs.

Patients accepting inclusion in the project will get specialised palliative care throughout their trajectory, within three weeks after diagnosis until end-of-life or cure without residual palliative care needs.

Both patients participating in the project and patients referred on-demand will receive four-weekly visits in their homes. Patients participating in the project are guaranteed that the first visit will take place within three weeks after diagnosis, whereas patients referred on-demand might have to wait longer before they meet the palliative care team.

ELIGIBILITY:
Inclusion Criteria:

* Adults newly diagnosed with pancreatic cancer in Dept. of Surgery, Hospital of North Zealand, Denmark
* Caregivers involved in care or practical help

Exclusion Criteria:

* Inability to take an active part in answering questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with pancreatic cancer in Dept. of Surgery, Hospital of North Zealand, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Use of healthcare services | Until death or end of study, an average of 8 months
  Number of acute hospital admissions and number of days in hospital

SECONDARY OUTCOMES:
Survival | Until death or end of study, an average of 8 months
  Survival
Quality of life: EORTC QLQ-C15-PAL | Four-weekly until death or end of study, an average of 8 months
  Quality of life measured using the questionnaire: EORTC QLQ-C15-PAL
Quality of life: EORTC QLQ-PAN26 | Four-weekly until death or end of study, an average of 8 months
  Quality of life measured using the questionnaire: EORTC QLQ-PAN26
Anxiety and/or depression | Four-weekly until death or end of study, an average of 8 months
  Anxiety and/or depression measured using the questionnaire: HADS
Change in weight | Four-weekly until death or end of study, an average of 8 months
  Weight in kilos
Preferred and actual place of death | Until death or end of study, an average of 8 months
  Advance care planning (where patients prefer to die) and the actual place of death
Carer satisfaction with palliative care | Three-monthly. The last time is at a follow-up visit after the patient has died, or at end of study, an average of 10 months
  Carer satisfaction with palliative care measured using the questionnaire: FAMCARE-2

CONTACTS AND LOCATIONS:
Overall Officials: Inge H Dufva, Principal Investigator — Consultant, Palliative Care Unit, Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Frederikssund, Denmark